CLINICAL TRIAL: NCT00360373
Title: Adolescent Gastric By-pass and Diabetic Precursors
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: DK68228; R03DK068228 (NIH)
Record Dates: First submitted 2006-08-02; First posted 2006-08-04 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2014-01

CONDITIONS: Obesity
Keywords: bariatric; obesity; insulin resistance; gastric bypass; adolescent
MeSH Terms: conditions — Obesity; Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this research study is to find out what effects (good and bad) gastric bypass has on metabolism, including pancreatic insulin secretion. In addition, we will compare the effects of gastric bypass on the metabolism of adults and adolescents to try to determine whether there are greater metabolic and health advantages of performing gastric bypass earlier in life versus waiting until adulthood.

DETAILED DESCRIPTION:
Overweight and obesity are the most common metabolic disorders affecting the U.S. with 31% of adults and 16% of adolescents now meeting Centers for Disease Control criteria for these conditions. As the obesity epidemic has unfolded, so too has the increase in prevalence of abnormalities of carbohydrate metabolism. The single most effective treatment for type 2 diabetes in severely obese adults may be bariatric surgery, a procedure that is most commonly performed in the 5th and 6th decades of life. While it is clear that rapid and profound weight loss can significantly improve carbohydrate metabolism in adults, it is not clear to what degree type 2 diabetes is reversible in these patients. The pathophysiology of type 2 diabetes in adolescents and children is not well understood and no studies have yet examined the effect of surgical weight loss on insulin resistance, insulin secretion, or glucose tolerance in severely obese young people. However, it seems likely that bariatric surgery could improve these conditions in youth. Understanding the relative benefits of surgically induced weight reduction on carbohydrate metabolism in adolescents compared to older subjects is important for determining optimal timing of this intervention. This knowledge may also lead to key insights into obesity-induced diabetes. In this project we will test the hypothesis that bariatric surgical intervention will more effectively improve insulin resistance, β cell dysfunction, and glucose tolerance in adolescents compared to adults. Three specific aims are proposed: 1) To compare the derangements of carbohydrate metabolism among very severely obese (body mass index ≥ 40 kg/m2) adolescents and adults referred for bariatric surgery; 2) To assess improvement in carbohydrate metabolism longitudinally (during and after surgical weight loss) comparing differences in the mechanisms of improvement between the two age groups; 3) To compare major complications in the two age groups following bariatric surgery. These data will provide critical information about age-related metabolic outcomes of bariatric surgery and could inform the design of larger studies to examine the role of early bariatric surgery in management of disorders related to insulin resistance in patients at high risk for these conditions.

ELIGIBILITY:
Inclusion Criteria:

* Approved to be scheduled for laparoscopic gastric bypass surgery for VSO at Cincinnati Children's or University Hospital
* Age at time of gastric bypass surgery date >15 and <21 years, or >30 and <45 years
* BMI >40
* Weight at age 18 consistent with severe adolescent obesity (if height < 5'5" weight > 200 pounds or if height >5'5", weight > 250)

Exclusion Criteria:

* Diagnosis of cirrhosis, total bilirubin >1 mg/dL, prothrombin time > 13.3 sec
* Prior myocardial infarction
* Serum creatinine >1.7mg/dL
* Systemic (PO, IV, IM) glucocorticoid therapy within the previous six weeks prior to blood sampling
* Peri-menopausal (irregularity of menstrual periods over the past 3 months (67) or demonstrated abnormally high follicle stimulating hormone levels (68)
* Severe T2DM (on insulin for control of hyperglycemia, or HbA1c > 8.5)

Ages: 15 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Adolescents undergoing weight loss surgery
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2005-08; Primary Completion 2009-03 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Insulin Resistance | 2 weeks, 3 months, and 12 months
  This study uses the frequently sampled intravenous glucose tolerance test (FSIVGTT) to determine the effects of bariatric surgery on insulin resistance, carbohydrate metabolism, β cell dysfunction, and glucose tolerance for this adolescent cohort. Carbohydrate metabolism will be assessed by measuring plasma glucose and insulin concentrations in blood samples obtained during fasting as well as during FSIVGTT at baseline and all subsequent time points..

CONTACTS AND LOCATIONS:
Overall Officials: Thomas H Inge, MD, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Result] Jeffreys RM, Hrovat K, Woo JG, Schmidt M, Inge TH, Xanthakos SA. Dietary assessment of adolescents undergoing laparoscopic Roux-en-Y gastric bypass surgery: macro- and micronutrient, fiber, and supplement intake. Surg Obes Relat Dis. 2012 May-Jun;8(3):331-6. doi: 10.1016/j.soard.2011.11.016. Epub 2011 Dec 10. PMID 22260884
- [Derived] Inge TH, Prigeon RL, Elder DA, Jenkins TM, Cohen RM, Xanthakos SA, Benoit SC, Dolan LM, Daniels SR, D'Alessio DA. Insulin Sensitivity and beta-Cell Function Improve after Gastric Bypass in Severely Obese Adolescents. J Pediatr. 2015 Nov;167(5):1042-8.e1. doi: 10.1016/j.jpeds.2015.08.020. Epub 2015 Sep 9. PMID 26363548